CLINICAL TRIAL: NCT04413409
Title: A Trial Evaluating the Efficacy of Metastasectomy in Patients With Oligo-Metastatic Breast Cancer
Brief Title: A Trial Evaluating the Efficacy of Metastasectomy in Patients With Oligo-Metastatic Breast Cancer(OMIT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Chief Physician, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUSCC-OMIT
Record Dates: First submitted 2020-03-07; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer
Keywords: metastasectomy; oligo-metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Metastasectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgical group (Experimental): The metastatic sites are firstly treated by surgery then followed by systemic treatment
  Interventions: Procedure: Metastasectomy for the metastatic sites
- systemic group (No Intervention): After confirmation of puncture, receive systemic treatment

INTERVENTIONS:
Procedure: Metastasectomy for the metastatic sites — patients randomized to this group will receive metastasectomy for the metastatic sites then followed by the systemic therapy
  Arms: surgical group

SUMMARY:
This is a randomized clinical trial (OMIT study) evaluating the efficacy of metastasectomy in patients with oligo-metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. women aged 18-70 years old;
2. ECOG score: 0-2 points;
3. the expected life period is more than 3 months;
4. Histologically confirmed metastatic breast cancer: locations include central lung lesions, peripheral lung lesions or liver metastases;
5. PET-CT or other imaging showed patients with ≤3 metastastatic sites, involving 1-2 organs mentioned above, single lesion ≤5cm;
6. according to the RECIST 1.1 edition, there is at least one measurable lesion;
7. the main organs are functioning normally, meeting the following criteria: Blood routine: Hb > 90g/L (no blood transfusion within 14 days); ANC > 1.5 x 109/L; PLT > 75 * 109/L;Liver function: total bilirubin TBIL is less than 1.5 x ULN (upper limit of normal value); ALT and AST are less than 3 x ULN; if there is liver metastasis, ALT and AST are less than 5 x ULN;Renal function: serum creatinine < 1 x ULN;
8. participants voluntarily joined the study, signed informed consent, and followed up.

Exclusion Criteria:

1. the number of metastastatic sites ≥ 3, or the surgeon determines that the R0 resection cannot be achieved;
2. with metastatic lesions other than liver or lung
3. patients with local recurrence
4. palliative radiation therapy or interventional therapy have been performed previously for metastatic lesions
5. has received systemic treatment for metastatic disease, such as chemotherapy, targeted therapy, endocrine therapy, immunotherapy, etc.
6. pregnant or lactating women, women of childbearing age who cannot practice effective contraceptives;
7. involvement in clinical trials of unlisted drugs within 4 weeks before the start of this study;
8. severe cardiopulmonary insufficiency, severe liver and kidney insufficiency;

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 172 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2023-03-10 (Estimated); Study Completion 2025-03-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 3-year
  Overall survival is calculated from randomization to death from any cause

SECONDARY OUTCOMES:
Time To Event (TTE) | From date of randomization at baseline to the time of the first event, assessed up to 60 months
  From date of randomization at baseline to the time of the first event (Disease progression, local recurrence or distant metastasis, contralateral breast cancer, second primary tumor, or death from any cause), whichever came first, assessed up to 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No